CLINICAL TRIAL: NCT02739230
Title: Comparing Pain Relief Between Exparel® Injection vs. On-Q Catheter as the Postsurgical Analgesia Following Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESmith2016
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis: Joint Replacement Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Exparel Injection (Active Comparator)
  Interventions: Drug: Exparel
- On-Q intraarthicual catheter placement (Active Comparator)
  Interventions: Drug: On-Q pain intra-articular catheter

INTERVENTIONS:
Drug: Exparel
  Arms: Exparel Injection
Drug: On-Q pain intra-articular catheter
  Arms: On-Q intraarthicual catheter placement

SUMMARY:
The goal of this research project is to evaluate the effectiveness of a novel treatment to control pain after Total Knee Arthroplasty (TKA). The proposed approach to manage pain and eliminate risks associated with catheters is the use of Exparel injection into the joint at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults scheduled to undergo primary total knee replacement
2. Willing and able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-12; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total Morphine and morphine equivalent consumption | 96 hours post-op